CLINICAL TRIAL: NCT05802927
Title: A Randomized Controlled Trial to Determine the Effects of Diabetes-specific Formula on Glycemic Control in Individuals With Type 2 Diabetes
Brief Title: Diabetes-specific Formula (DSF) in Individuals With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BL65
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Diabetes-specific formula (Other)
  Interventions: Other: DSF
- Experimental: Breakfast 1 Noodle Soup (Other)
  Interventions: Other: Breakfast 1
- Experimental: Breakfast 2 Glutinous rice (Other)
  Interventions: Other: Breakfast 2

INTERVENTIONS:
Other: DSF — Diabetes-specific formula
  Arms: Experimental: Diabetes-specific formula
Other: Breakfast 1 — Noodle Soup
  Arms: Experimental: Breakfast 1 Noodle Soup
Other: Breakfast 2 — Glutinous rice
  Arms: Experimental: Breakfast 2 Glutinous rice

SUMMARY:
A randomized, controlled, crossover design with three treatments to determine the effects of diabetes-specific formula on glycemic control in individuals with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Has type 2 diabetes as evidenced by use of oral antihyperglycemic medication(s).
2. BMI > 18.5 and ≤ 35.0 kg/m2.
3. Weight stable.
4. Male or non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit.
5. If on chronic medication, the dosage to be constant for at least two months prior to screening visit and to maintain the medication and dose throughout the study.
6. Willing to follow the protocol throughout the study.
7. At least a two-week washout period between completion of a previous research study and their start in the current study.
8. Willing to refrain from taking non-study diabetes-specific formulas over the course of the study.
9. Voluntarily signed and dated an Informed Consent Form (ICF) prior to any participation in the study.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

1. Has a screening HbA1c level < 7% or ≥ 10%.
2. Uses exogenous insulin for glucose control.
3. Has confirmed type 1 diabetes and/or had history of diabetic ketoacidosis.
4. Has current infection, inpatient surgery or received systemic corticosteroid treatment in the last 3 months; or received antibiotics in the last 3 weeks.
5. Has active malignancy.
6. Has significant cardiovascular event within 6 months prior to study entry or history of congestive heart failure.
7. Has end stage organ failure or was post organ transplant.
8. Has a history of renal disease or severe gastroparesis.
9. Has current hepatic disease.
10. Has had bariatric surgery including gastric balloon; history of gastrointestinal disease or intestinal surgery that can interfere with consumption or digestion or absorption of study product.
11. Has a chronic, contagious, infectious disease.
12. Has eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures.
13. Taking any herbals, dietary supplements or medications other than allowed anti-hyperglycemic medications, during the past four weeks prior to screening visit that could profoundly affect blood glucose or appetite.
14. Uses diabetes-specific formula(s) defined as more than one eating occasion per week in the last three months.
15. Has clotting or bleeding disorders.
16. Participates in another study that has not been approved as a concomitant study by Abbott Nutrition.
17. Has allergy or intolerance to any ingredient in the study product.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Postprandial blood glucose | 3 hours
  Positive area under the curve (AUC) for blood glucose concentration from 0 to 180 minutes.

SECONDARY OUTCOMES:
Postprandial insulin | 3 hours
  Positive area under the curve (AUC) for blood insulin concentration from 0 to 180 minutes.
Appetite | 3 hours
  Negative/Positive area under the curve (AUC) for each item of Appetite questionnaire from 0 to 180 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Siew Ling Tey, PhD, Study Chair — Abbott Nutrition R&D
Locations (2):
- Thailand (2):
  - Chulalongkorn University, Bangkok
  - Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No